CLINICAL TRIAL: NCT01961999
Title: "Early" and "Late" Timing Indication for Starting Renal Replacement Therapy in Acute Renal Failure After Cardiac Surgery: a Prospective, Controlled, Interventional, Single-center Trial
Brief Title: Early Versus Late Renal Replacement Therapy After Cardiac Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ospedali Riuniti Ancona (Other)
Responsible Party: Principal Investigator, Giuseppe Crescenzi M.D., Medical Doctor Cardiac Surgery intensive care Unit, Ospedali Riuniti Ancona
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ANCCH01
Record Dates: First submitted 2013-10-06; First posted 2013-10-14 (Estimated); Last update posted 2013-10-14 (Estimated); Status verified 2013-10

CONDITIONS: Acute Kidney Injury
Keywords: Acute kidney injury; Cardiac surgery; Renal replacement therapy
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Early RRT (Active Comparator): In the "early" arm renal replacement therapy was started on the basis of refractory oliguria: urine output <0,5ml/Kg/h for > 6 hours
  Interventions: Procedure: Early RRT
- Late RRT (Active Comparator): In the "late" arm at least one the following criteria must be fulfilled prior to initiation of renal replacement therapy:
  * persistent and refractory oliguria (<0,5 ml/Kg/h >12h), despite therapy
  * refractory extravascular fluid overload
  * azotemia > 40mmol/L or 240 mg/dL
  * metabolic acidosis (pH<7,2)
  * hyperkaliemia (k+>6 mmol/L)
  Interventions: Procedure: Late RRT

INTERVENTIONS:
Procedure: Early RRT — In the "early" arm renal replacement therapy was started on the basis of refractory oliguria: urine output <0,5ml/Kg/h for > 6 hours
  Arms: Early RRT
Procedure: Late RRT — In the "late" arm at least one the following criteria must be fulfilled prior to initiation of renal replacement therapy:
  persistent and refractory oliguria (<0,5ml/Kg/h >12h), despite therapy refractory extravascular fluid overload azotemia >40mmol/L or 240mg/dL metabolic acidosis (pH<7,2) hyperkaliemia (k+>6mmol/L)
  Arms: Late RRT

SUMMARY:
The question of timing of initiation of renal replacement therapy (RRT), "early" versus "late", has seldom been the focus of high-quality or rigorous evaluation. As a consequence, initiatives aimed at identifying the "optimal timing of initiation of RRT" in acute kidney injury (AKI) have been given the highest priority for investigation by the Acute Kidney Injury Network (AKIN). Accordingly, the investigators conducted a prospective, controlled, interventional trial, comparing two treatment groups in which the only variable was the RRT initiation strategy, to determine whether "early" versus "late" initiation in patients with AKI after cardiac surgery is associated with a survival benefit or more favorable outcomes.

DETAILED DESCRIPTION:
Acute kidney injury after cardiac surgery is strongly associated with in-hospital mortality and morbidity. This is an area where effective treatments are lacking and trial are difficult to perform. To date no randomized controlled trial (RCT) has sufficiently estimated the impact of RRT timing of initiation on patient outcome, and the present prospective, controlled, interventional, single-center trial attempts to compare patient outcome with "early" versus "late" initiation of RRT. Previous studies in cardiac surgery setting have been retrospective ones and have been hampered by lead-time bias, and drop out patients. To overcome these biases all patients who underwent cardiac surgery were prospectively enrolled in the trial and were divided in two treatment groups: the "early" approach was used during the first 10-months, and the "late" approach during the next 10-months. To improve the information gained from this non-classical randomized study and to minimize bias, the investigators enrolled almost all patients with few exclusion criteria during two following short periods, used intention-to-treat analysis and treated all patients according to local protocols and international guidelines, except for RRT initiation strategy.

Outcome parameters were hospital mortality, and ICU and hospital length of stay.

"Early" therapy was started after 6 hours of urine output of less than<0,5ml/Kg/h, whereas in the "late" group RRT therapy was started on the basis of persistent (lasting more than 12 hours) oliguria.

Data obtained from the database were analyzed using "Statistical Package for Social Science" (SPSS Inc, Chicago, IL). Continuous variables are presented as mean±SD, categorical variables were summarized as frequencies and percentages. The Student t test or Pearson X square test were performed to evaluate differences between groups and to analyze subgroups. For statistics, a p<0.05 was considered significant.

Power calculation was based on previous reports13 on cumulative mortality following cardiac surgery. 50% reduction of mortality was hypothesized when the more conservative approach to cardiac surgery-AKI was applied. The suggested number of patients was about 900 patients per group.

The main limitation of the present study include the non-classical randomization, nevertheless we conducted an interventional trial comparing two treatment strategies in two different groups of patients, prospectively followed and suitable for both treatments.

ELIGIBILITY:
Inclusion criteria:

* Patients submitted to cardiac surgery at "Ospedali Riuniti" of Ancona during the study period
* Planned use of extracorporeal circulation

Exclusion criteria:

* Preoperative dialysis
* Planned off-pump cardiac surgery
* Pts (or proxy) did not sign informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1800 (Actual)
Dates: Start 2011-07; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
operative mortality | death during the same hospitalization as surgery, or after discharge, but within 30 days of surgery
  death during the same hospitalization as surgery, or after discharge, but within 30 days of surgery

SECONDARY OUTCOMES:
Hospital length of stay | during the same hospitalization for surgery, but within 30 days from surgery
  Hospital length of stay (days): from operative day to discharge or death
ICU length of stay | during the same hospitalization for surgery, but within 30 days from surgery
  from entrance to ICU after the end of surgery to discharge to ward facilities

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Crescenzi, MD, Principal Investigator — Ospedali Riuniti di Ancona
Locations (1):
- Cardiac Surgery department of Ospedali Riuniti, Ancona, AN, Italy

REFERENCES:
- [Background] Karkouti K, Wijeysundera DN, Yau TM, Callum JL, Cheng DC, Crowther M, Dupuis JY, Fremes SE, Kent B, Laflamme C, Lamy A, Legare JF, Mazer CD, McCluskey SA, Rubens FD, Sawchuk C, Beattie WS. Acute kidney injury after cardiac surgery: focus on modifiable risk factors. Circulation. 2009 Feb 3;119(4):495-502. doi: 10.1161/CIRCULATIONAHA.108.786913. Epub 2009 Jan 19. PMID 19153273
- [Background] Bellomo R, Ronco C, Kellum JA, Mehta RL, Palevsky P; Acute Dialysis Quality Initiative workgroup. Acute renal failure - definition, outcome measures, animal models, fluid therapy and information technology needs: the Second International Consensus Conference of the Acute Dialysis Quality Initiative (ADQI) Group. Crit Care. 2004 Aug;8(4):R204-12. doi: 10.1186/cc2872. Epub 2004 May 24. PMID 15312219
- [Background] Gibney N, Hoste E, Burdmann EA, Bunchman T, Kher V, Viswanathan R, Mehta RL, Ronco C. Timing of initiation and discontinuation of renal replacement therapy in AKI: unanswered key questions. Clin J Am Soc Nephrol. 2008 May;3(3):876-80. doi: 10.2215/CJN.04871107. Epub 2008 Mar 5. PMID 18322044
- [Background] Chertow GM, Lazarus JM, Christiansen CL, Cook EF, Hammermeister KE, Grover F, Daley J. Preoperative renal risk stratification. Circulation. 1997 Feb 18;95(4):878-84. doi: 10.1161/01.cir.95.4.878. PMID 9054745
- [Background] Bouman CS, Oudemans-Van Straaten HM, Tijssen JG, Zandstra DF, Kesecioglu J. Effects of early high-volume continuous venovenous hemofiltration on survival and recovery of renal function in intensive care patients with acute renal failure: a prospective, randomized trial. Crit Care Med. 2002 Oct;30(10):2205-11. doi: 10.1097/00003246-200210000-00005. PMID 12394945
- [Background] Korevaar JC, Jansen MA, Dekker FW, Jager KJ, Boeschoten EW, Krediet RT, Bossuyt PM; Netherlands Cooperative Study on the Adequacy of Dialysis Study Group. When to initiate dialysis: effect of proposed US guidelines on survival. Lancet. 2001 Sep 29;358(9287):1046-50. doi: 10.1016/S0140-6736(01)06180-3. PMID 11589934
- [Background] Prowle JR, Bellomo R. Continuous renal replacement therapy: recent advances and future research. Nat Rev Nephrol. 2010 Sep;6(9):521-9. doi: 10.1038/nrneph.2010.100. Epub 2010 Jul 20. PMID 20644583
- [Background] Bagshaw SM, Gibney RT, McAlister FA, Bellomo R. The SPARK Study: a phase II randomized blinded controlled trial of the effect of furosemide in critically ill patients with early acute kidney injury. Trials. 2010 May 11;11:50. doi: 10.1186/1745-6215-11-50. PMID 20459801
- [Background] Akins CW, Miller DC, Turina MI, Kouchoukos NT, Blackstone EH, Grunkemeier GL, Takkenberg JJ, David TE, Butchart EG, Adams DH, Shahian DM, Hagl S, Mayer JE, Lytle BW; Councils of the American Association for Thoracic Surgery; Society of Thoracic Surgeons; European Assoication for Cardio-Thoracic Surgery; Ad Hoc Liaison Committee for Standardizing Definitions of Prosthetic Heart Valve Morbidity. Guidelines for reporting mortality and morbidity after cardiac valve interventions. J Thorac Cardiovasc Surg. 2008 Apr;135(4):732-8. doi: 10.1016/j.jtcvs.2007.12.002. No abstract available. PMID 18374749
- [Background] Kuitunen A, Vento A, Suojaranta-Ylinen R, Pettila V. Acute renal failure after cardiac surgery: evaluation of the RIFLE classification. Ann Thorac Surg. 2006 Feb;81(2):542-6. doi: 10.1016/j.athoracsur.2005.07.047. PMID 16427848
- [Background] Uchino S, Bellomo R, Goldsmith D, Bates S, Ronco C. An assessment of the RIFLE criteria for acute renal failure in hospitalized patients. Crit Care Med. 2006 Jul;34(7):1913-7. doi: 10.1097/01.CCM.0000224227.70642.4F. PMID 16715038
- [Background] Cooper WA, O'Brien SM, Thourani VH, Guyton RA, Bridges CR, Szczech LA, Petersen R, Peterson ED. Impact of renal dysfunction on outcomes of coronary artery bypass surgery: results from the Society of Thoracic Surgeons National Adult Cardiac Database. Circulation. 2006 Feb 28;113(8):1063-70. doi: 10.1161/CIRCULATIONAHA.105.580084. Epub 2006 Feb 20. PMID 16490821
- [Background] Pierri MD, Capestro F, Zingaro C, Torracca L. The changing face of cardiac surgery patients: an insight into a Mediterranean region. Eur J Cardiothorac Surg. 2010 Oct;38(4):407-13. doi: 10.1016/j.ejcts.2010.02.040. PMID 20399675
- [Background] Bove T, Calabro MG, Landoni G, Aletti G, Marino G, Crescenzi G, Rosica C, Zangrillo A. The incidence and risk of acute renal failure after cardiac surgery. J Cardiothorac Vasc Anesth. 2004 Aug;18(4):442-5. doi: 10.1053/j.jvca.2004.05.021. PMID 15365924
- [Background] Chertow GM, Levy EM, Hammermeister KE, Grover F, Daley J. Independent association between acute renal failure and mortality following cardiac surgery. Am J Med. 1998 Apr;104(4):343-8. doi: 10.1016/s0002-9343(98)00058-8. PMID 9576407
- [Background] Bagshaw SM, Uchino S, Bellomo R, Morimatsu H, Morgera S, Schetz M, Tan I, Bouman C, Macedo E, Gibney N, Tolwani A, Oudemans-van Straaten HM, Ronco C, Kellum JA; Beginning and Ending Supportive Therapy for the Kidney (BEST Kidney) Investigators. Timing of renal replacement therapy and clinical outcomes in critically ill patients with severe acute kidney injury. J Crit Care. 2009 Mar;24(1):129-40. doi: 10.1016/j.jcrc.2007.12.017. Epub 2008 Apr 18. PMID 19272549
- [Background] Pannu N, Klarenbach S, Wiebe N, Manns B, Tonelli M; Alberta Kidney Disease Network. Renal replacement therapy in patients with acute renal failure: a systematic review. JAMA. 2008 Feb 20;299(7):793-805. doi: 10.1001/jama.299.7.793. PMID 18285591
- [Background] Liu KD, Himmelfarb J, Paganini E, Ikizler TA, Soroko SH, Mehta RL, Chertow GM. Timing of initiation of dialysis in critically ill patients with acute kidney injury. Clin J Am Soc Nephrol. 2006 Sep;1(5):915-9. doi: 10.2215/CJN.01430406. Epub 2006 Jul 6. PMID 17699307
- [Background] Metnitz PG, Krenn CG, Steltzer H, Lang T, Ploder J, Lenz K, Le Gall JR, Druml W. Effect of acute renal failure requiring renal replacement therapy on outcome in critically ill patients. Crit Care Med. 2002 Sep;30(9):2051-8. doi: 10.1097/00003246-200209000-00016. PMID 12352040
- [Background] Ympa YP, Sakr Y, Reinhart K, Vincent JL. Has mortality from acute renal failure decreased? A systematic review of the literature. Am J Med. 2005 Aug;118(8):827-32. doi: 10.1016/j.amjmed.2005.01.069. PMID 16084171
- [Background] Kellum JA. Acute kidney injury. Crit Care Med. 2008 Apr;36(4 Suppl):S141-5. doi: 10.1097/CCM.0b013e318168c4a4. PMID 18382185
- [Derived] Crescenzi G, Torracca L, Pierri MD, Rosica C, Munch C, Capestro F. 'Early' and 'late' timing for renal replacement therapy in acute kidney injury after cardiac surgery: a prospective, interventional, controlled, single-centre trial. Interact Cardiovasc Thorac Surg. 2015 May;20(5):616-21. doi: 10.1093/icvts/ivv025. Epub 2015 Feb 18. PMID 25694207